CLINICAL TRIAL: NCT03214133
Title: Determining an Optimal Dose of Epicatechin-Rich Chocolate and Its Effect on Performance
Brief Title: Effects of Epicatechin-rich Cocoa on Collagen Synthesis
Acronym: coca-dose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1020494
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Collagen Synthesis

STUDY DESIGN:
Intervention Model Description: Arm 1 of the project will employ a randomized single-blinded crossover design with subjects completing all 4 of the epicatechin-rich chocolate trials (0, 1, 2 and 3 mg.kg-1). Arm 2 will use a randomized parallel double-blind design with neither the subjects nor the investigators knowing who is on which treatment (optimized epicatechin-rich chocolate dose or Dutch processed/epicatechin depleted placebo.
Who Masked: Participant, Investigator
Masking Description: Alkalized (0.01 mg epicatechin/g) ) and non alkalized cocoa (4.1 mg epicatechin/g) will be mixed in various ratios to achieve the desired 0, 1, 2, 3 mg/ kg body mass but maintaining equally weighed dose of cocoa for each intervention.
  For Arm 2, the same quantity of either alkalized or non alkalized cocoa will be given to achieve the optimized dosed of epicatechin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epicatechin Dose Response (Experimental): This arm will investigate varying doses of epicatechin on procollagen type I N-terminal propeptide (PINP) at varying doses CON, 1, 2, 3 mg/kg body mass.
  Interventions: Other: Epicatechin-rich cocoa dose response
- Epicatechin-rich cocoa on performance (Placebo Comparator): Athletes will ingest the optimized dose of epicatechin-rich cocoa vs placebo alongside maximum power training to determine if this nutritional intervention results in a greater increase in RFD and performance than maximum power training alone.
  Interventions: Other: Epicatechin-rich cocoa vs placebo on performance

INTERVENTIONS:
Other: Epicatechin-rich cocoa dose response — Subjects consume randomized doses of 0, 1, 2, 3 mg epicatechin/kg from epicatechin-rich cocoa. The optimal dose of epicatechin-rich chocolate will be the dose which have the greatest increase PNIP levels.
  Arms: Epicatechin Dose Response
Other: Epicatechin-rich cocoa vs placebo on performance — An optimized dose of epicatechin-rich cocoa or placebo will be given for 3 weeks alongside a prescribed power-based training program. In a randomized parallel design the effect of the optimal dose of epicatechin-rich chocolate, compared to placebo, on maximal isometric squat force, RFD, and jump testing will be quantified.
  Arms: Epicatechin-rich cocoa on performance

SUMMARY:
This study will investigate the effects of dietary supplementation of epicatechin-rich cocoa in humans on collagen synthesis and power-based performance outcomes (rate of force development).

DETAILED DESCRIPTION:
The investigators have recently completed a study looking at the expression of the collagens following consumption of increasing doses of epicatechin in rats . This data clearly shows that increasing doses of epicatechin, either 0.5 mg.kg-1 delivered once, twice, or three times a day, or 2 mg.kg-1 once a day, results in increasing expression of the fibrillar collagens (I, III, and V). This preliminary data suggests that epicatechin-rich chocolate supplementation can increase collagen expression in humans and that this may improve force transfer. From this background, the hypothesis proposed is that supplementation with epicatechin-rich chocolate will increase rate of force development and performance in athletes. Therefore, this simple nutrition intervention has the potential to simultaneously improve performance, decrease injuries and accelerate return to competition through improved collagen synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Collegiate level male athletes between the ages of 18¬-25 years of age, currently participating in sport, will be recruited to participate in the study.

Exclusion Criteria:

* History of more than 3 musculoskeletal injuries within the past 12 months.
* Health and dietary restriction (e.g. lactose intolerance) that would be affected by the supplementation protocol.
* The initial phase will be performed in males since collagen synthesis varies significantly throughout the menstrual cycle in females. Since collagen synthesis is the main outcome measure for the study this would confound the initial phase of the work. Provided this work proves successful then the investigators will aim to proceed with similar research in females.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Epicatechin-rich cocoa dose response | ~26 days
  investigating effects doses of 0, 1, 2, 3 mg epicatechin/kg/day procollagen type I N-terminal propeptide (PINP) in the blood after 5 days of supplementation with 2-day wash out between.
Effect of the optimized dose of epicatechin-rich cocoa on performance | ~22 days
  Performance measures (of rate of force development) will be quantified for 3 weeks alongside the ingestion of an optimized dose of epicatechin-rich cocoa vs placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Baar, PhD, Principal Investigator — UC Davis
Locations (1):
- Neurobiology, Physiology & Behaviour, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be made available to other researchers. Any data shared will be published in a blinded manner.